CLINICAL TRIAL: NCT00769080
Title: A Prospective, Multicentre, Controlled, Observational Study to Evaluate the Performance of Patient Support Programme (PSP) in Improving Patient Adherence With Adjuvant Aromatase Inhibitors (AI) Medication for Postmenopausal, Early Stage Breast Cancer
Brief Title: The Performance of Patient Support Program in Early Stage Breast Cancer
Acronym: ARI NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCN-ARI-2008/1
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: PSP; Standard Treatment; Standard Treatment plus PSP
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Standard Treatment plus PSP
- 2: Standard Treatment

SUMMARY:
The purpose of this study is to compare the 1-year adherence to upfront adjuvant AI for postmenopausal, early stage breast cancer in the two observational arms; Standard Treatment and Standard Treatment plus PSP arm after one year

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated written Informed Consent
* Have been taking upfront AI adjuvant therapy in line with current SmPC
* Be capable of completing drug intake by herself
* Be capable of understanding Chinese

Exclusion Criteria:

* Upfront adjuvant hormonal therapy by an AI to which upfront adjuvant indication has not been granted by SFDA
* Upfront adjuvant AI medication which has exceeded over eight weeks
* Previous adjuvant hormonal therapy for breast cancer lasting over 8 weeks other than AI
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with hormone sensitive early breast cancers to whom have been prescribed upfront adjuvant AI medication (aromatase inhibitors; anastrozole or letrozole) according to the current product SmPC. The upfront AI medication must not have exceeded eight weeks.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2008-09; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
compare the 1-year adherence | 1 year

SECONDARY OUTCOMES:
scores of Beliefs about Medicines Questionnaire (BMQ) | 1 year
Scores in Patient Centred Care Questionnaire (PCCQ) | 1 year
Morisky scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — AstraZeneca; Emily Huang, Study Chair — AstraZeneca; Shen Zhenzhou, Prof, Principal Investigator — Fudan University
Locations (13):
- China (13):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Harbin, Heilongjiang
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Yu KD, Zhou Y, Liu GY, Li B, He PQ, Zhang HW, Lou LH, Wang XJ, Wang S, Tang JH, Liu YH, Wang X, Jiang ZF, Ma LW, Gu L, Cao MZ, Zhang QY, Wang SM, Su FX, Zheng H, Li HY, Tang LL, Sun SR, Liu JP, Shao ZM, Shen ZZ. A prospective, multicenter, controlled, observational study to evaluate the efficacy of a patient support program in improving patients' persistence to adjuvant aromatase inhibitor medication for postmenopausal, early stage breast cancer. Breast Cancer Res Treat. 2012 Jul;134(1):307-13. doi: 10.1007/s10549-012-2059-8. Epub 2012 Apr 12. PMID 22527106